CLINICAL TRIAL: NCT05843422
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of Single and Multiple Topical Doses of QY211 Gel in Healthy Chinese Subjects and Patients With Mild to Moderate Atopic Dermatitis
Brief Title: A First-in-Human Study of QY211 Gel in Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: E-nitiate Biopharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QY211-Ⅰ-1
Record Dates: First submitted 2023-03-06; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- part 1-0.8% QY211 Gel or placebo（10%BSA） (Experimental): 6 subjects use 0.8% QY211 Gel，2 subject uses 0.8% QY211 placebo ，11days（Day1 QD,Day4-Day10 BID,Day11 QD ）.
  Interventions: Drug: 0.8% QY211 Gel or placebo
- part 1-1.5% QY211 Gel or placebo（10%BSA） (Experimental): 6 subjects use 0.8% QY211 Gel，2 subject uses 0.8% QY211 placebo ，11days（Day1 QD,Day4-Day10 BID,Day11 QD ）.
  Interventions: Drug: 1.5% QY211 Gel or placebo
- part 1-1.5% QY211 Gel or placebo（20%BSA） (Experimental): 6 subjects use 0.8% QY211 Gel，2 subject uses 0.8% QY211 placebo ，11days（Day1 QD,Day4-D10 BID,Day11 QD ）.
  Interventions: Drug: 1.5% QY211 Gel or placebo
- part 2-0.1% QY211 Gel or placebo (Experimental): 6 subjects use 0.1% QY211 Gel，2 subject uses 0.1% QY211 placebo ，29days（Day1-Day28 BID,Day29 QD）.
  Interventions: Drug: 0.1% QY211 Gel or placebo
- part 2-0.3% QY211 Gel or placebo (Experimental): 6 subjects use 0.3% QY211 Gel，2 subject uses 0.3% QY211 placebo ，29days（Day1-Day28 BID,Day29 QD）.
  Interventions: Drug: 0.3% QY211 Gel or placebo
- part 2-0.8% QY211 Gel or placebo (Experimental): 6 subjects use 0.3% QY211 Gel，2 subject uses 0.3% QY211 placebo ，29days（Day1-Day28 BID,Day29 QD）.
  Interventions: Drug: 0.8% QY211 Gel or placebo
- part 2-1.5% QY211 Gel or placebo (Experimental): 6 subjects use 0.3% QY211 Gel，2 subject uses 0.3% QY211 placebo ，29days（Day1-Day28 BID,Day29 QD）.
  Interventions: Drug: 1.5% QY211 Gel or placebo

INTERVENTIONS:
Drug: 0.1% QY211 Gel or placebo — QY211 Gel or placebo topical applied to skin
  Arms: part 2-0.1% QY211 Gel or placebo
Drug: 0.3% QY211 Gel or placebo — QY211 Gel or placebo topical applied to skin
  Arms: part 2-0.3% QY211 Gel or placebo
Drug: 0.8% QY211 Gel or placebo — QY211 Gel or placebo topical applied to skin
  Arms: part 1-0.8% QY211 Gel or placebo（10%BSA）; part 2-0.8% QY211 Gel or placebo
Drug: 1.5% QY211 Gel or placebo — QY211 Gel or placebo topical applied to skin
  Arms: part 1-1.5% QY211 Gel or placebo（10%BSA）; part 1-1.5% QY211 Gel or placebo（20%BSA）; part 2-1.5% QY211 Gel or placebo

SUMMARY:
This is a phase Ia/Ib,Randomized, Double-Blind, Placebo-Controlled Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of Single and Multiple Topical Doses of QY211 Gel in Healthy Chinese Subjects and Patients with Mild to Moderate Atopic Dermatitis

ELIGIBILITY:
Inclusion Criteria:

Part 1

1. Male or female subjects (male or female) aged 18-45 years (inclusive);
2. Body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females; body mass index (BMI) within the range of 18.0 to 27.0 kg/m2 (including the cut-off value);
3. the investigator determined vital signs, physical examination, clinical laboratory test values (blood routine, urine routine, blood biochemistry, coagulation function, pregnancy test (female), hepatitis, HIV, syphilis), routine 12-lead ECG results in line with healthy subjects
4. the subject fully understood the purpose, nature, methods and possible adverse reactions of the trial, volunteered to participate, and signed informed consent before the start of any study procedures;
5. the subject was able to communicate well with the investigator, and understand and comply with the requirements of this study.

Part 2

1. Male and female patients aged 18-65 years (including the boundary value);
2. Meet Hanifin-Rajka diagnostic criteria at screening and have a history of AD for at least 6 months ;
3. IGA score of 2 (mild) or 3 (moderate) at screening and baseline;
4. The total area of atopic dermatitis lesions is 5% -20% BSA
5. Patients fully understand the purpose, nature, methods and possible adverse reactions of the trial, voluntarily participate, and sign an informed consent form before the start of any study procedures;
6. Patients can communicate well with the investigator and comply with the study and follow-up procedures;

Exclusion Criteria:

Part 1

1. Allergic constitution, such as allergic to two or more drugs and food; or known to be allergic to the composition of this drug (QY201 and excipients: carbomer (homopolymer type B 974P NF), edetate disodium, sodium hydroxide, propylene glycol and purified water);
2. Patients who have received surgery within 3 months before screening, or plan to undergo surgery during the study period, or have received surgery that will affect drug absorption, distribution, metabolism and excretion;
3. Previous or current cardiovascular, liver, kidney, respiratory, blood and lymphatic, endocrine, immune, mental, neurological, gastrointestinal system, metabolism and bone diseases, and the investigators believe that the subjects have clinical significance, not suitable for the trial;
4. Patients who can not tolerate venipuncture, have a history of fainting needle, halo blood;
5. History or presence of clinically relevant skin diseases that, in the opinion of the investigator, contraindicate the study or affect the assessment of the site of administration, including psoriasis, eczema, acne, atopic dermatitis, dysplastic mole, other skin lesions, history of skin cancer, or skin diseases that affect the safety evaluation of the test drug;
6. Vaccination with live (attenuated) vaccines within 2 months prior to screening;
7. Smoking or drinking within 3 months before screening (smoking: > 10 cigarettes/day; drinking: > 15 g pure alcohol/day, equivalent to 450 mL beer, 150 mL wine or 50 mL low-grade liquor), or alcohol and drug abuse (morphine/methylamphetamine/ketamine/methylenedioxyamphetamine/tetrahydrocannabinolic acid/cocaine) test positive;
8. Participated in other drug or device clinical trials within 3 months before screening;
9. Non-physiological blood loss ≥ 400 mL (including trauma, blood collection, blood donation) within 3 months before screening, or plan to donate blood during the study or within 1 month after the end of the study;
10. Pregnant women, lactating women, or subjects who have plans to donate sperm or eggs, or (including male and female subjects) refuse to voluntarily take effective contraceptive measures from the screening period to 6 months after the end of the last dose;
11. Use of any other drugs, including oral or topical drugs such as prescription drugs, over-the-counter drugs, and herbal medicines, except vitamins and/or paracetamol, within 2 weeks before screening;
12. Drinking excessive tea, coffee and/or caffeine-rich beverages (more than 8 cups, 1 cup = 250 mL) every day within 3 months before screening;
13. Subjects have skin conditions in the target application area (back, lateral arm area) that affect the tolerability assessment of the study, such as tattoos;
14. Subjects who are judged unsuitable for participation by other investigators;

Part 2

1. Patients with or suspected active tuberculosis, latent untreated tuberculosis, incompletely cured tuberculosis or Mycobacterium tuberculosis infection (except for treatment records that prove that patients have been adequately treated, according to the medical judgment of the investigator and/or infectious disease experts, can enter this study) as judged by the investigator and/or infectious disease specialist (combined with medical history, symptoms, signs, laboratory tests, T-spot test, imaging examination);
2. Hepatitis B surface antigen (HBsAg) positive or hepatitis C virus antibody (HCV-Ab) positive during screening; or HIV antibody or Treponema pallidum antibody positive;
3. Patients with any clinical symptoms of bacterial, viral, parasitic or fungal infection requiring treatment during the screening period;
4. Previous disseminated herpes zoster (single attack), or disseminated herpes simplex (single attack), or recurrent (≥ 2 attacks) local herpes zoster;
5. Patients with a history of mental illness or genetic history of mental illness or epilepsy, the use of antipsychotic drugs, sedative drugs;
6. In addition to a history of atopic dermatitis, previous history of other connective tissue diseases, or severe cardiovascular, liver, kidney, digestive tract, nerve, skin and other diseases, or patients with malignant tumors (except completely removed cervical carcinoma in situ or non-metastatic cutaneous squamous cell carcinoma or basal cell carcinoma), systemic sex hormone therapy or other interventions may be required, and participation in this study may be at risk as judged by the investigator;
7. Patients with non-immune factors (such as hyperlipidemia, diabetes, thyroid disease, severe heart abnormalities, etc.);
8. Patients who have previously suffered from lymphatic diseases, or have signs or symptoms of lymphoproliferative diseases, including but not limited to lymph nodes or splenomegaly;
9. In addition to atopic dermatitis, suffering from other skin diseases that affect the evaluation of the test results, or the presence of large tattoos, birthmarks, skin scars and other conditions in the skin lesions;
10. Known immunodeficiency disease or first-degree relatives with hereditary immunodeficiency disease;
11. Patients with cerebral hemorrhage or cerebral infarction within 1 year;
12. Patients with previous thromboembolism (including deep venous thrombosis, pulmonary embolism, arterial thrombosis, etc.) or other high-risk groups prone to thromboembolism;
13. Previous or planned organ transplantation (such as liver and kidney transplantation);
14. Clinical or laboratory tests judged by the investigator as abnormal with clinical significance;
15. History of alcoholism or drug abuse within 6 months before screening;
16. Participated in any investigational drug 4 weeks (or 5 half-lives, whichever is longer) before screening or participated in any medical device clinical trial within 3 months;
17. Non-physiological blood loss ≥ 400 mL (including trauma, blood sampling, blood donation) within 3 months before screening, or plan to donate blood during the study or within 1 month after the end of the study;
18. Patients with the following cardiac abnormalities:

    1. Acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting or coronary stent implantation within 3 months prior to screening;
    2. Severe arrhythmia (e.g., second-degree type 2 or third-degree atrioventricular block, long QT syndrome or QTcF abnormalities: male > 470 ms female > 480 ms, atrial fibrillation, frequent premature beats);
    3. Decompensated cardiac insufficiency (NYHA class III or IV);
    4. Other cardiac diseases requiring treatment and assessed by the investigator as inappropriate for participation in this study;
19. Systemic or local use of JAK inhibitors (eg, Ruxolitinib, Tofacitinib, Baricitinib, Filgotinib, Lestaurtinib, Pacritinib, Delgocitinib, Upadacitinib, Abrocitinib, etc) within 3 months prior to screening;
20. Major surgical procedures or serious trauma within 8 weeks prior to screening or anticipation of major surgical procedures during the trial (defined as major surgical procedures referring to Grade 3 and 4 procedures as specified in the Measures for the Management of Clinical Applications of Medical Technology implemented on November 1, 2018), and all surgical or major trauma-related AEs had not recovered (recovered to CTCAEv5.0 ≤ Grade 1 or baseline) before screening.
21. Received biological therapy for atopic dermatitis (including but not limited to dupilumab) within 8 weeks (or 5 elimination half-lives, whichever is longer) before randomization;
22. Received live (attenuated) vaccine within 4 weeks before randomization, or planned to receive live (attenuated) vaccine during treatment and within 4 weeks after the last use of investigational product;
23. Patients who have used long-acting anticoagulants (such as warfarin, dabigatran, etc.) or need to continue anticoagulant therapy (except aspirin ≤ 100 mg/day) within 4 weeks before randomization;
24. Receiving systemic therapy (including glucocorticoids, cyclosporine, mycophenolate mofetil, interferon γ, azathioprine, methotrexate, tripterygium wilfordii tablets and other Chinese herbal medicines) known or likely to affect atopic dermatitis within 4 weeks (or 5 half-lives, whichever is longer) before randomization, phototherapy (such as UVB, PUVA, etc.) or receiving antihistamines within 2 weeks before randomization;
25. Patients who have received topical drugs known or likely to affect atopic dermatitis within 2 weeks before randomization, including but not limited to topical glucocorticoids (TCS), calcineurin inhibitors (TCI), topical phosphodiesterase 4 (PDE 4) inhibitors;
26. Use of topical antibiotics, antibacterial soap, sodium hypochlorite in the target application area within 7 days before randomization, or use of emollients not provided by the sponsor or designated by the investigator within 12 hours before baseline;
27. Allergic constitution or suspected allergy to the active ingredients or excipients of the investigational drug;
28. Pregnant women, lactating women, or patients (including male and female patients) refuse to voluntarily take effective contraceptive measures during the screening period until 6 months after the end of the last dose (see Appendix 2 for details);
29. Do not avoid prolonged exposure to natural or artificial ultraviolet (UV) radiation, or plan to perform such exposure during the study, and the investigator believes that it may affect atopic dermatitis;
30. Any patient considered unsuitable for participation in this clinical study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-23 (Estimated); Study Completion 2024-10-23 (Estimated)

PRIMARY OUTCOMES:
Part1:Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 to Day 13
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part1:Number of Participants With Clinical Laboratory Abnormalities | Day 3 to Day 13
  A treatment-emergent laboratory abnormality was defined as an increase of at least 1 abnormality grade from baseline and occurring after the first dose of study drug
Part1:Number of Participants With Clinically Significant Changes Form Baseline in Physical Examination | Day 3 to Day 13
Part1:Number of Participants With Clinically Significant Treatment-emergent Electrocardiogram (ECG) Findings | Day 3 to Day 13
  ECG data will be monitored
Part 1:Number of Participants With Clinically Significant Changes Form Baseline in Vital Signs | Day 1 to Day 13
Part 1:Severity of local skin irritation | Day 1 to Day 13
  Skin irritation response assessment recording method: ① subjective symptoms: including itching, pain, or burning sensation, evaluated according to the 4-level method: 0=none; 1=mild, without affecting daily life and sleep; 2=Moderate, affecting daily life but not sleep; 3=Severe, affecting sleep.The signs of skin lesions include erythema, papules, edema, blisters, bullae, exudates, pustules, erosion, exudates, ulcers, hypertrophy, desquamation, etc., which can be evaluated according to the 4-level method: 0=none; 1=Mild, with only blurred erythema, no edema (skin lesions not palpable), and papules; 2=Moderate, clear erythema with edema (skin lesions can be touched) and papules; "3=Severe, with blisters, bullae, exudates or pustules, erosion, exudates or ulcers.
Part 2:Number of Participants With Adverse Events (AEs) and Serious Adverse Events | Day 1 to Day 31
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part2:Number of Participants With Clinical Laboratory Abnormalities | Day 8 to Day 29
  A treatment-emergent laboratory abnormality was defined as an increase of at least 1 abnormality grade from baseline and occurring after the first dose of study drug
Part2:Number of Participants With Clinically Significant Changes Form Baseline in Physical Examination | Day 8 to Day 29
Part2:Number of Participants With Clinically Significant Treatment-emergent Electrocardiogram (ECG) Findings | Day 8 to Day 29.
  ECG data will be monitored
Part 2:Number of Participants With Clinically Significant Changes Form Baseline in Vital Signs | Day 8 to Day 30

SECONDARY OUTCOMES:
Rate of change from baseline in Eczema Area and Severity Index (EASI) in patients（part 2 only） | Up to 4 weeks
  EASI quantifies severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema, induration /papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs ) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.
Proportion of patients with at least a 2-point improvement in IGA score from baseline（part 2 only） | Up to 4 weeks
  The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participants' psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).Proportion of patients with Investigator's Global Assessment (IGA) score of 0 or 1 and an improvement of at least 2 points in IGA score from baseline at 1, 2, 3 and 4 weeks after treatment.
Percentage of Participants Achieving >=50%/75%/90% Improvement From Baseline in Eczema Area and Severity Index (EASI-50/EASI-75/EASI-90) Response（part2 only） | Up to 4 weeks
  EASI quantifies severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema, induration/papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs ) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.
Change from baseline in Peak daily Pruritus NRS score (PP-NRS) （part 2 only） | Up to 29 days
  Change from baseline in Peak daily Pruritus NRS score (PP-NRS) during treatment.Using a 0 to 10 point scale, 0 represents "" no itching "" and 10 represents "" worst itch imaginable ""，Rating the degree of itchiness experienced in the past 24 hours.
Rate of change from baseline in SCORAD score （part 2 only） | Up to 4 weeks
  SCORAD (Severity Scoring of Atopic Dermatitis) Change from Baseline to Week 8 of atopic dermatitis lesion as measured by the Scoring of Atopic Dermatitis (SCORAD). SCORAD is a composite severity index comprising a) the amount/extent of body area affected; b) 2 subjective symptom of pruritus (0-10 points) and sleep disturbance measured (0-10 points); and c) 6 disease intensity assessments [Dryness/Scaling, Erythema, Excoriation, Induration/Papulation, Lichenification and Oozing/ Weeping/Crusting, each grades from 0 (None) to 3 (Severe). A SCORAD score ranges from 0 (No AD present) to 103.
Change from baseline in total score of Dermal Quality of Life Index Questionnaire (DLQI) （part 2 only） | Up to 4 weeks
  The DLQI is a dermatology-specific quality of life (QOL) instrument designed to assess impact of disease on a participants QOL. It is a 10-item questionnaire that, in addition to evaluating overall, QOL can be used to assess 6 different aspects: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships and treatment. Questions scored on a 4-point Likert scale: 0 (not relevant), 1 (a little), 2 (a lot), and 3 (very much). Scores of individual items (0-3) were added to yield a total score (0-30); higher score = greater impairment of participants QOL.
Rate of change from baseline in atopic dermatitis in BSA（part 2 only） | Up to 4 weeks
  Rate of change from baseline in atopic dermatitis in BSA at Weeks 1, 2, 3, and 4 postdose.
Tmax of QY211-Single and Multiple Dose Drugs | Up to 29 days
  Time of maximum concentration(single Dose and Steady state PK)
Cmax of QY211-Single and Multiple Dose Drugs | Up to 29 days
  Maximum observed plasma concentration(single Dose and Steady state PK)
t1/2 of QY211-Single and Multiple Dose Drugs | Up to 29 days
  The time it takes for the blood concentration of the drug to drop by half from the highest value in the body(single Dose and Steady state PK)
AUC QY211-Single and Multiple Dose Drugs | Up to 29 days
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration(single Dose and Steady state PK)

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No